CLINICAL TRIAL: NCT02460627
Title: Postoperative Pain Management With Topical Lidocaine After Arthroscopy on Knee. A Randomized Double-blind Study
Brief Title: Topical Lidocaine After Arthroscopy on Knee
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20150006
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Pain; Topical Anaesthesia
Keywords: Arthroscopy; Meniscus; Lidocaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Surgical Tape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine adhesive tape (Experimental)
  Interventions: Drug: Lidocaine adhesive tape
- Adhesive tape (Placebo Comparator)
  Interventions: Other: Adhesive tape

INTERVENTIONS:
Drug: Lidocaine adhesive tape — 700 mg for 12 hours
  Arms: Lidocaine adhesive tape
Other: Adhesive tape — For 12 hours
  Arms: Adhesive tape

SUMMARY:
More than half of the patients suffer from intensive pain 1-2 days after arthroscopy in the knee. Walking function and physical activities are affected by this intensive pain although local anaesthetic is given in the joint and soft tissue.

The patients are often discharged on the same day as the arthroscopy takes place depending on their ability to walk with or without assistive technology.

It is a well-known fact that the patient is given a dose of morphine, analgesics or an ice pack on a painful knee to reduce pain intensity. The aim of the project is to study whether pain intensity and analgesics can be additionally reduced by giving local anaesthetic by means of an adhesive tape placed on the skin instead of giving morphine, analgesics or ice pack on a painful knee.

The researchers plan to include a cohort of 180 patients: 60 patients having a meniscus sutured, 60 patients having meniscus tissue removed surgically, 60 patients having mucous fold removed surgically.

This study is planned to be a pilot study in order to complete a future large medical science study.

ELIGIBILITY:
Inclusion Criteria:

* Planned resection of meniscus (DS832, DM232)
* Planned meniscus suture (DS832)
* Planned plica resection (DM659)
* Patients >=18 years and <50 years
* Statement of consent
* Tolerance to Lidocaine (analgesics)

Exclusion Criteria:

* Type 1 diabetes or type 2 diabetes
* Allergic to Lidocaine (analgesics)
* Heart disease, liver disease, kidney disease
* BMI >=35
* Unability to read or speak Danish
* Rheumatoid arthritis or other degenerative diseases in joint, bone structure or cartilage
* Insufficient coagulation
* Medication of morphine pre-operatively
* Pregnant and nursing women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Administration of analgesics or morphine in time | 1 day
  First time administration of analgesics or morphine in time on demand

SECONDARY OUTCOMES:
Discharges of patients in time | 1 day
Value Added Score (VAS) estimation of pain | 1 day
  Estimate pain at each administration of analgesics on demand before discharge of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Region of Northern Jutland, Denmark